CLINICAL TRIAL: NCT02748863
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, 52-weeks Study to Demonstrate the Efficacy, Safety and Tolerability of Subcutaneous Secukinumab Injections With 2 mL Pre-filled Syringes (300 mg) in Adult Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Study of Secukinumab With 2 mL Pre-filled Syringes
Acronym: ALLURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2323
Record Dates: First submitted 2016-03-08; First posted 2016-04-22 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Psoriasis
Keywords: psoriasis; secukinumab; pre-filled syringes
MeSH Terms: conditions — Psoriasis | interventions — secukinumab; Metabolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo, provided in a 2 mL pre-filled syringe Placebo, provided in a 1 mL pre-filled syringe
  Interventions: Drug: Placebo
- Secukinumab 2 mL form (Experimental): Secukinumab 300 mg, provided in a 2 mL pre-filled syringe
  Interventions: Drug: Secukinumab 2 mL form
- Secukinumab 1 mL form (Active Comparator): Secukinumab 300 mg provided in 2 pre-filled syringes of 1 mL/150 mg (current approved form)
  Interventions: Drug: Secukinumab 1 mL form

INTERVENTIONS:
Drug: Placebo — 2 mL + 2 x 1 mL Placebo s.c. at randomization, weeks 1, 3, and 4, thereafter 4-weekly until week 48
  Arms: Placebo
Drug: Secukinumab 2 mL form — Secukinumab 300 mg/2mL + 2 x 1 mL placebo s.c. at randomization, week 1 , 3, 4, thereafter 4-weekly until Week 48
  Arms: Secukinumab 2 mL form
Drug: Secukinumab 1 mL form — Secukinumab 150 mg/1mL x 2 + 2 mL placebo s.c. at randomization, week 1 , 3, 4, thereafter 4-weekly until Week 48
  Arms: Secukinumab 1 mL form

SUMMARY:
The aim of the study was to demonstrate efficacy, safety and tolerability of 2 mL pre-filled syringe of 300 mg secukinumab in treatment of moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a 52-weeks multicenter, randomized, double-blind, placebo-controlled, parallel-group trial in 24 subjects with moderate to severe plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for inclusion in this study must fulfill all of the following criteria:

1. Subjects must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study related activity is performed. Where relevant, a legal representative will also sign the informed study consent according to local laws and regulations.
2. Men or women of at least 18 years of age at the time of Screening.
3. Chronic plaque-type psoriasis present for at least 6 months and diagnosed before Randomization.
4. Moderate to severe psoriasis as defined at Randomization by:

   * PASI score of 12 or greater, and
   * IGA mod 2011 score of 3 or greater (based on a scale of 0 - 4), and
   * Body Surface Area (BSA) affected by plaque-type psoriasis of 10% or greater.
5. Candidate for systemic therapy. This is defined as a subject having moderate to severe chronic plaque-type psoriasis that is inadequately controlled by

   * Topical treatment and/or
   * Phototherapy and/or
   * Previous systemic therapy

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis) at Screening or Randomization.
2. Ongoing use of prohibited treatments. Washout periods detailed in the protocol have to be adhered to. Subjects not willing to limit UV light exposure (e.g., sunbathing and/or the use of tanning devices) during the course of the study will be considered not eligible for this study since UV light exposure is prohibited.

   Note: administration of live vaccines 6 weeks prior to Randomization or during the study period is also prohibited.
3. Previous exposure to secukinumab (AIN457) or any other biologic drug directly targeting IL-17 or the IL-17 receptor.
4. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days until the expected pharmacodynamic effect has returned to baseline, whichever is longer; or longer if required by local regulations.
5. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
6. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system treated or untreated within the past 5 years, regardless of whether there is evidence of local recurrence or metastases (except for Bowen's disease, or basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 12 weeks; carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
7. History of hypersensitivity to any of study drug constituent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2018-06-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (14):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Fountain Valley, California
  - Novartis Investigative Site, Fremont, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, Saint Joseph, Missouri
  - Novartis Investigative Site, Verona, New Jersey
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Sugar Land, Texas
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Tacoma, Washington
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Liège
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Surrey, British Columbia
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, München
- Novartis Investigative Site, Kopavogur, Iceland
- Latvia (5):
  - Novartis Investigative Site, Daugavpils, LVA
  - Novartis Investigative Site, Jelgava, LVA
  - Novartis Investigative Site, Riga, LVA
  - Novartis Investigative Site, Ventspils, LVA
  - Novartis Investigative Site, Riga
- Poland (2):
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Warsaw
- Russia (4):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (7):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sant Joan Despí, Barcelona
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Pontevedra
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Bursa
  - Novartis Investigative Site, Izmir
- United Kingdom (4):
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Dundee
  - Novartis Investigative Site, Surrey

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sigurgeirsson B, Schakel K, Hong CH, Effendy I, Placek W, Rich P, Keefe D, Bruin G, Charef P, Fu R, Hampele I, Patekar M. Efficacy, tolerability, patient usability, and satisfaction with a 2 mL pre-filled syringe containing secukinumab 300 mg in patients with moderate to severe plaque psoriasis: results from the phase 3 randomized, double-blind, placebo-controlled ALLURE study. J Dermatolog Treat. 2022 May;33(3):1718-1726. doi: 10.1080/09546634.2021.1902925. Epub 2021 Apr 26. PMID 33896356

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 251 patients were screened and 214 patients were randomized
Groups:
- Secukinumab 2 mL PFS: Secukinumab 300 mg in one 2 mL pre-filled syringe
- Secukinumab 2 x 1 mL PFS: Secukinumab 300 mg provided in 2 pre-filled syringes of 1 mL/150 mg (current approved form)
- Secukinumab 2 mL PFS Following Placebo: Switched from placebo to secukinumab 300 mg, provided in one 2 mL pre-filled syringe
- Secukinumab 2 x 1 mL PFS Following Placebo: Switched from placebo to secukinumab 300 mg provided in 2 pre-filled syringes of 1 mL/150 mg
Period: Treatment Period 1
Arm/Group | Secukinumab 2 mL PFS | Secukinumab 2 x 1 mL PFS | Placebo | Secukinumab 2 mL PFS Following Placebo | Secukinumab 2 x 1 mL PFS Following Placebo
Started | 72 | 71 | 71 | 0 (Not applicable for this period) | 0 (Not applicable for this period)
Completed | 72 | 69 | 69 | 0 | 0
Not Completed | 0 | 2 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0
Period: Treatment Period 2
Arm/Group | Secukinumab 2 mL PFS | Secukinumab 2 x 1 mL PFS | Placebo | Secukinumab 2 mL PFS Following Placebo | Secukinumab 2 x 1 mL PFS Following Placebo
Started | 72 | 69 | 0 | 34 | 34
Completed | 67 | 66 | 0 | 32 | 33
Not Completed | 5 | 3 | 0 | 2 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 2 mL PFS | Secukinumab 2 x 1 mL PFS | Placebo | Total
Number analyzed (Participants) | 72 | 71 | 71 | 214
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 68 | 64 | 68 | 200
  >=65 years | 4 | 7 | 3 | 14
  >=75 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 25 | 81
  Male | 44 | 43 | 46 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 64 | 64 | 66 | 194
  Black | 2 | 1 | 1 | 4
  Asian | 4 | 4 | 4 | 12
  Pacific Islander | 0 | 1 | 0 | 1
  Other | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Participants With Psoriasis Area and Severity Index (PASI) 75 Response After 12 Weeks of Treatment
Description: Number of participants who achieved ≥ 75% reduction in PASI compared to baseline
  PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: 12 weeks
Population: The full analysis set (FAS) population was used for this analysis. The FAS included all participants to whom treatment was assigned. Only participants from the FAS, who had values at a given week, were included in the analysis for that week.
Measure: Number; unit: participants
Groups:
- Placebo: Placebo, in a 2 mL pre-filled syringe Placebo, in a 1 mL pre-filled syringe
Arm/Group | Secukinumab 2 mL PFS | Placebo
Number analyzed (Participants) | 72 | 71
participants | 64 | 1
Statistical Analysis 1: Comparison: Secukinumab 2 mL PFS vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 717.42, 95% CI 2-sided [68.00 to 7569.56]

2. Secondary Outcome: Participants With PASI 90 After 12 Weeks of Treatment
Description: Number of participants who achieved ≥ 90% and 100% reduction in PASI compared to baseline
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Secukinumab 2 mL PFS | Placebo
Number analyzed (Participants) | 72 | 71
participants | 48 | 1
Statistical Analysis 1: Comparison: Secukinumab 2 mL PFS vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 168.39, 95% CI 2-sided [21.20 to 1337.22]

3. Secondary Outcome: Number of Participants With PASI 100 Response After 12 Weeks of Treatment
Description: Participants who achieved 100% reduction in PASI compared to baseline
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Secukinumab 2 mL PFS | Secukinumab 2 x 1 mL PFS | Placebo
Number analyzed (Participants) | 72 | 71 | 71
participants | 28 | 26 | 0
Statistical Analysis 1: Comparison: Secukinumab 2 mL PFS vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided; Risk Difference (RD) = 38.75, 95% CI 2-sided [27.41 to 50.09]
Statistical Analysis 2: Comparison: Secukinumab 2 x 1 mL PFS vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided; Risk Difference (RD) = 36.48, 95% CI 2-sided [25.19 to 47.76]

4. Secondary Outcome: Number of Participants Achieving PASI 50/75/90/100 Response or IGA 0 or 1 Response
Description: PASI response over time up to week 52: Number of participants who achieved ≥ 50%, 75%, 90% and 100% reduction in PASI and achieve IGA mod 2011 0 or 1 and improved by at least 2 points on the IGA scale compared to baseline
Time Frame: up to week 52
Population: FAS
Measure: Number; unit: participants
Groups:
- Placebo: Placebo, in a 2 mL pre-filled syringe Placebo, in a 1 mL pre-filled syringe
  From week 16 on is zero for all parameters in placebo group
Arm/Group | Secukinumab 2 mL PFS | Secukinumab 2 x 1 mL PFS | Placebo | Secukinumab 2 mL PFS Following Placebo | Secukinumab 2 x 1 mL PFS Following Placebo
Number analyzed (Participants) | 72 | 71 | 71 | 34 | 34
participants
  Week 1 IGA 0/1 | 1 | 0 | 0 | 0 | 0
  Week 1 PASI 50 | 5 | 5 | 1 | 0 | 1
  Week 1 PASI 75 | 0 | 2 | 0 | 0 | 0
  Week 1 PASI 90 | 0 | 0 | 0 | 0 | 0
  Week 1 PASI 100 | 0 | 0 | 0 | 0 | 0
  Week 2 IGA 0/1 | 2 | 1 | 1 | 0 | 1
  Week 2 PASI 50 | 18 | 28 | 1 | 1 | 0
  Week 2 PASI 75 | 4 | 5 | 0 | 0 | 0
  Week 2 PASI 90 | 0 | 1 | 0 | 0 | 0
  Week 2 PASI 100 | 0 | 1 | 0 | 0 | 0
  Week 3 IGA 0/1 | 6 | 11 | 1 | 0 | 1
  Week 3 PASI 50 | 39 | 40 | 5 | 3 | 1
  Week 3 PASI 75 | 14 | 17 | 0 | 0 | 0
  Week 3 PASI 90 | 4 | 4 | 0 | 0 | 0
  Week 3 PASI 100 | 0 | 1 | 0 | 0 | 0
  Week 4 IGA 0/1 | 19 | 23 | 0 | 0 | 0
  Week 4 PASI 50 | 53 | 52 | 6 | 5 | 1
  Week 4 PASI 75 | 29 | 32 | 1 | 1 | 0
  Week 4 PASI 90 | 10 | 13 | 0 | 0 | 0
  Week 4 PASI 100 | 3 | 3 | 0 | 0 | 0
  Week 8 IGA 0/1 | 43 | 41 | 0 | 0 | 0
  Week 8 PASI 50 | 66 | 60 | 5 | 3 | 2
  Week 8 PASI 75 | 53 | 51 | 0 | 0 | 0
  Week 8 PASI 90 | 35 | 31 | 0 | 0 | 0
  Week 8 PASI 100 | 8 | 11 | 0 | 0 | 0
  Week 12 IGA 0/1 | 55 | 49 | 1 | 0 | 0
  Week 12 PASI 50 | 67 | 61 | 5 | 2 | 2
  Week 12 PASI 75 | 64 | 58 | 1 | 0 | 0
  Week 12 PASI 90 | 48 | 50 | 1 | 0 | 0
  Week 12 PASI 100 | 28 | 26 | 0 | 0 | 0
  Week 16 IGA 0/1 | 57 | 52 | 0 | 14 | 5
  Week 16 PASI 50 | 69 | 61 | 0 | 27 | 20
  Week 16 PASI 75 | 65 | 60 | 0 | 17 | 13
  Week 16 PASI 90 | 56 | 55 | 0 | 8 | 4
  Week 16 PASI 100 | 37 | 31 | 0 | 5 | 1
  Week 28 IGA 0/1 | 64 | 54 | 0 | 30 | 25
  Week 28 PASI 50 | 71 | 66 | 0 | 33 | 30
  Week 28 PASI 75 | 69 | 60 | 0 | 32 | 28
  Week 28 PASI 90 | 62 | 56 | 0 | 26 | 21
  Week 28 PASI 100 | 44 | 34 | 0 | 16 | 12
  Week 40 IGA 0/1 | 60 | 55 | 0 | 28 | 25
  Week 40 PASI 50 | 69 | 67 | 0 | 33 | 33
  Week 40 PASI 75 | 66 | 63 | 0 | 31 | 31
  Week 40 PASI 90 | 58 | 57 | 0 | 27 | 24
  Week 40 PASI 100 | 40 | 37 | 0 | 20 | 17
  Week 52 IGA 0/1 | 55 | 55 | 0 | 28 | 26
  Week 52 PASI 50 | 67 | 67 | 0 | 31 | 32
  Week 52 PASI 75 | 63 | 62 | 0 | 30 | 31
  Week 52 PASI 90 | 54 | 58 | 0 | 25 | 26
  Week 52 PASI 100 | 40 | 37 | 0 | 20 | 16

5. Primary Outcome: Participants With IGA Mod 2011 0 or 1 After 12 Weeks of Treatment
Description: The Investigator's Global Assessment (IGA) mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. Treatment success was defined as achievement of IGA mod 2001 score of 0 or 1.
  Number of participants who achieved IGA mod 2011 0 or 1 and improved by at least 2 points on the IGA scale compared to baseline
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Secukinumab 2 mL PFS | Placebo
Number analyzed (Participants) | 72 | 71
participants | 55 | 1
Statistical Analysis 1: Comparison: Secukinumab 2 mL PFS vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 400.58, 95% CI 2-sided [47.48 to 3379.99]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for approximately 52 weeks. All cause mortality (deaths) was collected from First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV) up to a maximum of 52 weeks
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 52 weeks
Groups:
- Secukinumab 300 mg (2mL PFS): Treatment period 1 secukinumab 300 mg (2mL pre-filled syringes)
- AIN457 300 mg (2x1mL PFS): Treatment period 1 Secukinumab 300 mg in one 2 mL pre-filled syringe
- Placebo: Treatment period 1 Placebo
- Any AIN457 300 mg (2mL PFS): Any AIN457 300 mg (2 mL pre-filled syringes)
- Any Secukuinumab 300 mg (2x1mL PFS): Any AIN457 300 mg (2x1mL pre-filed syringes)
- Any Secukinumab 300 mg: Entire Any AIN457 300 mg
Arm/Group | Secukinumab 300 mg (2mL PFS) | AIN457 300 mg (2x1mL PFS) | Placebo | Any AIN457 300 mg (2mL PFS) | Any Secukuinumab 300 mg (2x1mL PFS) | Any Secukinumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/71 | 0/71 | 0/106 | 0/105 | 0/211
Serious Adverse Events (participants affected / at risk) | 0/72 | 1/71 | 2/71 | 8/106 | 5/105 | 13/211
Other Adverse Events (participants affected / at risk) | 33/72 | 39/71 | 29/71 | 60/106 | 68/105 | 128/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (2mL PFS) (N=72) | AIN457 300 mg (2x1mL PFS) (N=71) | Placebo (N=71) | Any AIN457 300 mg (2mL PFS) (N=106) | Any Secukuinumab 300 mg (2x1mL PFS) (N=105) | Any Secukinumab 300 mg (N=211)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 2
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (2mL PFS) (N=72) | AIN457 300 mg (2x1mL PFS) (N=71) | Placebo (N=71) | Any AIN457 300 mg (2mL PFS) (N=106) | Any Secukuinumab 300 mg (2x1mL PFS) (N=105) | Any Secukinumab 300 mg (N=211)
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 0 | 6 | 6 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 2 | 4
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 3 | 3 | 6
Toothache (Gastrointestinal disorders) | 2 | 0 | 2 | 3 | 1 | 4
Fatigue (General disorders) | 2 | 0 | 1 | 6 | 3 | 9
Injection site bruising (General disorders) | 2 | 1 | 1 | 2 | 2 | 4
Injection site erythema (General disorders) | 0 | 0 | 1 | 3 | 0 | 3
Injection site pruritus (General disorders) | 2 | 0 | 0 | 2 | 0 | 2
Injection site swelling (General disorders) | 0 | 2 | 0 | 0 | 2 | 2
Pyrexia (General disorders) | 2 | 1 | 0 | 2 | 2 | 4
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 1 | 2 | 3
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 3 | 2 | 5
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 2 | 4 | 6
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 3 | 3
Influenza (Infections and infestations) | 0 | 1 | 0 | 2 | 8 | 10
Nasopharyngitis (Infections and infestations) | 7 | 8 | 8 | 13 | 17 | 30
Oral herpes (Infections and infestations) | 3 | 0 | 2 | 3 | 3 | 6
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 5 | 1 | 6
Respiratory tract infection viral (Infections and infestations) | 2 | 0 | 1 | 2 | 5 | 7
Rhinitis (Infections and infestations) | 1 | 1 | 1 | 4 | 5 | 9
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 1 | 2 | 3
Tonsillitis (Infections and infestations) | 0 | 2 | 0 | 2 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 5 | 5 | 10
Vulvovaginal candidiasis (Infections and infestations) | 0 | 2 | 0 | 0 | 2 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1 | 3 | 4
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 3
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2 | 2 | 2 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 1 | 2
Weight increased (Investigations) | 2 | 0 | 0 | 3 | 0 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3 | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 6 | 4 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3 | 1 | 4
Headache (Nervous system disorders) | 6 | 6 | 3 | 10 | 8 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 4 | 3 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 4 | 1 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2 | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 3 | 10 | 4 | 14
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 3 | 3
Hypertension (Vascular disorders) | 0 | 1 | 3 | 3 | 5 | 8

LIMITATIONS AND CAVEATS:
"Other pre-specified outcomes" such as assess the subject usability and assessment of Dermatology Life Quality Index (DLQI) scores are exploratory in nature and are not reported in these results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT02748863/SAP_000.pdf
  • Study Protocol (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT02748863/Prot_001.pdf